CLINICAL TRIAL: NCT01971398
Title: Development of Education Materials for Prevention of Fetal Alcohol Syndrome (FAS) in Russia
Brief Title: Development of Education Materials for Prevention of FAS in Russia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTO1 2005-999-01
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Fetal Alcohol Spectrum Disorders; Fetal Alcohol Syndrome (FAS); Alcohol Related Neurodevelopmental Disorder; Alcohol Use Complicating Pregnancy, Unspecified Trimester
Keywords: Fetal Alcohol Spectrum Disorders (FASD); Prevention; Alcohol-Exposed Pregnancy; Knowledge; Attitudes
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Positive Brochure (Experimental): Women receive a "positive" FASD education brochure with positive images and are asked to read this brochure in the presence of a data collector.
  Interventions: Behavioral: Positive FASD education brochure
- Negative Brochure (Experimental): Women receive a "negative" FASD education brochure with negative, vivid images and are asked to read this brochure in the presence of a data collector.
  Interventions: Behavioral: Negative FASD education brochure
- A general women's health brochure (Active Comparator): Women receive a brochure on general aspects of women's health and pregnancy that is available in the Russian language and are asked to read this brochure in the presence of a data collector.
  Interventions: Behavioral: Active comparator (a general women's health brochure)

INTERVENTIONS:
Behavioral: Positive FASD education brochure — Exposure to a positive FASD education brochure
  Arms: Positive Brochure
Behavioral: Negative FASD education brochure — Exposure to a negative FASD education brochure
  Arms: Negative Brochure
Behavioral: Active comparator (a general women's health brochure) — Exposure to a general women's health brochure
  Arms: A general women's health brochure

SUMMARY:
This study is designed to increase knowledge and awareness to prevent Fetal Alcohol Syndrome in Russian children through development of printed FAS education materials targeting women of childbearing age in Russia. Alcohol abuse is a major public health problem in Russia. The rates of FAS and Alcohol Related Neurodevelopmental Disorders (ARND) in Russia are not precisely known. At this time, there are no programs to prevent FAS in Russia. The results of our previous study, focus groups with health professionals, pregnant women and their partners, non-pregnant women, and women with alcohol dependency, indicated limited knowledge about FAS, misconceptions about alcohol use during pregnancy, and a lack of materials and print resources related to this topic. Based on the initial findings, this proposal aims to develop and evaluate in a clinical trial informational brochures for women to increase knowledge and reduce drinking during pregnancy in Russia. The main hypotheses to be tested are:

* 1. Compared to the control group (CG) of women who receive a standard locally available flyer with health recommendations, women in the experimental groups who are exposed to printed information on FAS will show significantly more knowledge about FAS, significantly less acceptance of any alcohol use during pregnancy, and reduced drinking at one month follow-up assessment.
* 2. The group exposed to a brochure with negative images (IGN - Intervention group with a "negative brochure") regarding drinking during pregnancy will show significantly greater change in the predicted directions compared to the group exposed to positive images (IGP - Intervention group with a "positive" brochure) at the one month follow-up assessment.

DETAILED DESCRIPTION:
The study utilizes a randomized controlled trial design to test the two types of brochures (with positive vs. negative images and statements) to determine if either approach has more effect on women's alcohol consumption.

Pregnant and non-pregnant childbearing age women will be recruited at women's clinics and randomly assigned to participate in one of three groups: (1) participants will review the brochures that present information on FAS and alcohol use in pregnancy with positive images, (2) participants will review the brochures that that present information on FAS and alcohol use in pregnancy with negative, vivid images, and (3) participants will receive a general health information material that is available at their local clinics.

All study participants will complete a baseline survey assessing their attitudes toward drinking during pregnancy, knowledge of FAS, and current alcohol use. After that, the intervention will be conducted. The women in the two experimental groups will receive a brochure with either positive (IGP) or negative (IGN) images. The women will be asked to read one of two brochures in the presence of the data collector. If the participants ask questions, the data collector will redirect the participants to material in the brochure. Following the intervention, the women in the experimental groups will complete a brief questionnaire to assess their emotional responses to the materials and perceived effects. The women assigned to the control group (CG) will be asked to read a brochure on general aspects of women's' health. At a one-month follow-up, women in all three groups will complete a post-test of self-reported alcohol consumption, knowledge about prenatal effects of alcohol and FAS, and attitudes to drinking during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Childbearing age (between 18 and 44 years of age)
* Sexually active (any intercourse with a partner in the last year)
* Consume alcohol (any level of alcohol consumption in the last year)

Exclusion Criteria:

* None

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 422 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Changes in knowledge about Fetal Alcohol Syndrome (FAS) from baseline | 1 month follow-up
  A survey measure assessed knowledge about FAS
Changes in attitudes from baseline | 1 month follow-up
  A survey measure assessed attitudes and health beliefs related to alcohol use during pregnancy
Changes in alcohol consumption from baseline | 1 month follow-up
  Interviews assessed self-reported quantity/frequency of alcohol consumption and frequency of binge drinking and a detailed alcohol consumption report was received utilizing the Time Line Follow Back (TLFB) measure.

SECONDARY OUTCOMES:
Responses to brochures | After the intervention (reading an information brochure)
  A brief questionnaire to assess women's feedback, perceived effect, and emotional responses to health or FAS education brochures.

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Balachova, PhD, Principal Investigator — University of Oklahoma; Barbara Bonner, PhD, Principal Investigator — University of Oklahoma
Locations (3):
- University of Oklahoma, Oklahoma City, Oklahoma, United States
- Russia (2):
  - Nizhny Novgorod State Pedagogical University, Nizhny Novgorod
  - St. Petersburg State University, Saint Peterburg